CLINICAL TRIAL: NCT06770777
Title: Development And Evaluation of An Adaptive Web-Based Intervention for Whole Health Support For Patients With Chronic Pulmonology Obstructive Disease (COPD)
Brief Title: Development And Evaluation of An Adaptive Web-Based Intervention for COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-2639
Record Dates: First submitted 2024-12-30; First posted 2025-01-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-01

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: asynchronous; whole health support; website based intervention; implementation; access to whole health care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Psychotherapy

STUDY DESIGN:
Masking Description: Participants will choose which tier of the intervention that they are interested in accessing. Care providers will be notified about which services are accessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant led tiered intervention (Experimental): Participants living with COPD will navigate to the website and choose the tiered intervention that fits their needs. The first tier is information about COPD only. Second tier is reflective writing prompts for illness narrative generation and the third tier is asynchronous mental health support from a licensed clinical social worker.
  Interventions: Behavioral: Tiered whole health support for people living with COPD

INTERVENTIONS:
Behavioral: Tiered whole health support for people living with COPD — The website design allows study participants to choose the intervention tier(s) that meets their needs. There are three tiers from Tier 1: Information only, Tier 2 Reflective Writing, and Tier 3 LCSW Psychotherapeutic Intervention. Participants will also be able to choose multiple tiers if they are interested in continuing their participation. First Tier: The website offers standardized information about COPD care, healthcare navigation, and whole-person care. Information includes symptom management, disease progression and trajectory, healthcare navigation concepts, and directs people to the VA website with information about whole-person care. Second Tier: If participants choose, they can also select writing prompts with opportunities to reflect on their whole-person care and adjustment to illness. Third Tier: People living with COPD can also select to have asynchronous interaction with a licensed clinical social worker providing the narrative-based psychotherapeutic intervention.
  Other Names: Reflective writing prompts; Psychotherapy; Healthcare navigation and coaching

SUMMARY:
Narrative-based tiered asynchronous psychosocial and behavioral whole health support for people adjusting to living with COPD. The intervention is administered by experienced LCSWs under the PI's supervision.

DETAILED DESCRIPTION:
This study will advance health access equity for people with Chronic Obstructive Pulmonary Disease (COPD) by providing an asynchronous, patient-led, web-based, adaptive, flexible, and tiered intervention that easily integrates into the daily lives of both providers and patients living with COPD. This intervention includes health navigation education, health and behavior coaching, and narrative, strengths-based mental and behavioral health support. COPD is a complex chronic illness with multiple domains to study whole person support. Not only because of the significant impact of a lack of whole person support for people living with COPD but also because COPD shares many of the same symptomology and impact on daily living as other significant chronic illnesses such as heart failure, some neurological disorders, and some types of cancer (5-7). The lessons learned from studying COPD whole person support can be applied to other similar symptomatic burdensome chronic illnesses that also suffer from fragmented care.

ELIGIBILITY:
Inclusion Criteria:

* Has access to the internet once per week
* Has been diagnosed with COPD and is being seen at the ECHCS VA Medical Center or the University of Colorado Pulmonology clinics

Exclusion Criteria:

* Not in a conflicting research study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Personal Health Questionnaire- 9 item (PHQ9) | 0 months, 3 months
  The PHQ9 is a standardized, validated measurement used to track depression in both clinical and research settings.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 items (GAD7) | 0 months, 3 months
  The GAD7 is an established, validated measurement of anxiety in clinical and research settings.

OTHER OUTCOMES:
St George Respiratory Questionnaire (SGRQ) | 0 months, 3 months
  The SGRQ is an established and validated respiratory distress measurement for people with COPD in both clinical and research settings.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided